CLINICAL TRIAL: NCT01501890
Title: The Impact of Progesterone Treatment on Obstetrical Outcome Among Women With First Trimester Vaginal Bleeding
Brief Title: Progesterone for First Trimester Vaginal Bleeding
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: never started
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Adi Weintraub, Principal Investigator, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: sor003411ctil
Record Dates: First submitted 2011-09-09; First posted 2011-12-30 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Threatened Abortion; Pre-Eclampsia; Abruptio Placentae; Fetal Growth Retardation; Premature Birth
Keywords: Threatened Abortion; Progesterone; Subchorionic Hematoma; Pre-Eclampsia; Abruptio Placentae; Fetal Growth Retardation; Premature Birth
MeSH Terms: conditions — Abortion, Threatened; Pre-Eclampsia; Abruptio Placentae; Fetal Growth Retardation; Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Progesterone (Active Comparator): Women attending the Gynecological Emergency Unit due to first trimester vaginal bleeding, with a viable singleton pregnancy at a gestational age of 6-13 completed weeks of gestation
  Interventions: Drug: dihydroxyprogesterone caproate
- Placebo (Placebo Comparator): Women attending the Gynecological Emergency Unit due to first trimester vaginal bleeding, with a viable singleton pregnancy at a gestational age of 6-13 completed weeks of gestation.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: dihydroxyprogesterone caproate — 250mg once a week by intramuscular administration
  Other Names: 17a-Hydroxyprogesterone caproate
  Arms: Progesterone
Drug: Placebo — 0.9% NaCl
  Other Names: Sailine, Physiological water
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate whether treatment with progesterone for patients with first trimester vaginal bleeding will alter the rates of obstetrical complications and adverse pregnancy outcomes.

DETAILED DESCRIPTION:
First trimester vaginal bleeding is one of the most common pregnancy complications affecting 15-25% of all pregnancies. Threatened abortion is defined as bleeding through a closed cervical os in the first half of pregnancy. A subchorionic hematoma (SCH) is found in 18-39% of women with a threatened miscarriage and around 70% of women with a SCH will experience vaginal bleeding. Data on the relationship between first trimester vaginal bleeding and obstetric outcome is described mainly in retrospective and noncontrolled studies. It is hypothesized that first trimester bleeding is an indicator of a general tendency for complications (such as: preterm premature rupture of membranes (PPROM), preterm delivery (< 37 weeks gestation; PTD) low birth weight (<1500g; LBW) neonates, small for gestational age (SGA) neonates, placenta previa, placental abruption and stillbirth) later on in pregnancy.

Nowadays, there are not scientific based treatments for the prevention of complications associated with SCH and vaginal bleeding. Nevertheless, recent data have suggested that prophylactic administration of progesterone leads to a significant reduction in the rate of preterm deliveries and SGA neonates among patients with PTD or SGA neonates in the past. Although progesterone administration for threatened miscarriage was not studied, many physicians treat patients with first trimester vaginal bleeding with progesterone. In this era of evidence based medicine, the researchers aim to investigate whether treatment with progesterone for patients with first trimester vaginal bleeding will alter the rates of obstetrical complications and adverse pregnancy outcomes. The researchers hypothesize that treatment with progesterone for first trimester vaginal bleeding will alter the rates of the above mentioned obstetrical complications and adverse pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Low risk pregnancies
* Intrauterine pregnancy documented sonographically
* Singleton pregnancy
* Known gestational age
* Healthy women

Exclusion Criteria:

* Women after reproductive assistant techniques
* Women treated with progesterone
* Multiple pregnancies

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
adverse pregnancy outcomes | 9 months
  Miscarriage (also gestational age of miscarriage) Sonographic Intrauterine hematoma IUGR Placenta previa Pregnancy induced hypertension and preeclampsia/eclampsia Gestational age at delivery - Preterm delivery (before 37w); Early Preterm delivery (before 34w); and very early (before 28w) Mode of delivery Placental abruption PPROM Induction of labor PPH Apgar score Umbilical cord blood PH at birth Birth weight Fetal malformations Perinatal mortality Admission to the neonatal unit

SECONDARY OUTCOMES:
Uterine artery blood flow velocimetry | One month after recruitment upon completion of treatment
  Systolic to diastolic ratio, pulsatility index, resistance index and peak systolic velocity
Placental pathological examination | After delivey participants will be followed for the duration of hospital stay, an expected average of 3 days
  Placental weight and presence of infarcts, calcifications, fibrin deposits or signs of inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Ralika Hershkovitch, MD, Principal Investigator — Soroka University Medical Center
Locations (1):
- Soroka University Medical Center, Beersheba, Israel

REFERENCES:
- [Background] Lykke JA, Dideriksen KL, Lidegaard O, Langhoff-Roos J. First-trimester vaginal bleeding and complications later in pregnancy. Obstet Gynecol. 2010 May;115(5):935-944. doi: 10.1097/AOG.0b013e3181da8d38. PMID 20410766